CLINICAL TRIAL: NCT00158041
Title: Open-Label Prospective Trial Evaluating the Toxicities Associated With Subcutaneous Administration of Ethyol (Amifostine) for the Prevention of Radiation-Induced Toxicities
Brief Title: Subcutaneous Amifostine Safety Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mt. Sinai Medical Center, Miami (Other)
Collaborators: MedImmune LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ETH056-01D
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Head and Neck Cancer; Lung Cancer; Lymphoma
Keywords: Amifostine; Mucositis; Nausea; Hypotension; Rash
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Lymphoma; Mucositis; Nausea; Hypotension; Exanthema

INTERVENTIONS:
Drug: Amifostine administered subcutaneously

SUMMARY:
Amifostine is a radioprotective drug which is approved by the US FDA for administration prior to each radiation treatment using the intravenous route. The study evaluated the safety of amifostine administered subcutaneously. The four targeted toxicities were nausea/vomiting, hypotension, generalized skin rash, and injection-site skin reactions.

ELIGIBILITY:
Inclusion Criteria:

* Institutional criteria for administration of amifostine
* Radiation therapy
* ECOG PS of at least 2
* No distant mets
* Granulocyte count greater than 2000
* Platelet count greater than 100,000
* Creatinine less than 2.0

Exclusion Criteria:

* Allergy to amifostine
* Life expectancy less than 6 mos
* Investigational drug within last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452
Dates: Start 2002-01; Study Completion 2005-01

PRIMARY OUTCOMES:
Incidence of nausea/vomiting
Incidence of hypotension
Incidence of generalized skin rash
Incidence of injection-site skin toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Samuels, MD, Principal Investigator — Mt. Sinai Medical Center
Locations (1):
- Mt. Sinai Medical Center, Miami Beach, Florida, United States